CLINICAL TRIAL: NCT00035698
Title: Epidemiological and Genetic Studies of Body Mass Index
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-24244; R01HL068891 (NIH)
Record Dates: First submitted 2002-05-04; First posted 2002-05-06 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Diseases; Obesity; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — This study ended years ago, I do not know why I am being asked to update it as a clinical trial. It was never a clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify genes involved in obesity.

DETAILED DESCRIPTION:
BACKGROUND:

Increased levels of body mass index (BMI) are associated with increased mortality and morbidity from cardiovascular disease, hypertension, diabetes and other disorders. The frequency of obesity and its associated health-related problems is increasing in the American population.

DESIGN NARRATIVE:

The study builds upon a two-stage genome scan for BMI performed in the NHLBI Family Heart Study (FHS). In the first, 101 pedigrees were examined with 1027 persons genotyped and a LOD of 2.2 was found on chromosome 7. In stage 2, 135 sibships of 380 persons were examined , and a LOD of 3.2 was found for the same locus. Compelling linkage was found in the combined study (LOD = 4.9, chr 7q31.3, 137cM). The LOD or logarithm of odds is a statistical estimate of whether two loci (the sites of genes) are likely to lie near each other on a chromosome and are therefore likely to be inherited together as a package.

A novel strategy will be used which combines three cutting edge methods: (1) Regression Tree analyses to identify a homogenous subset of families with evidence for BMI linkage to 7q31.3; (2) DNA pooling of samples from linked versus unlinked families; and (3) quantitative PCR of DNA pools for very high-density single nucleotide polymorphism (SNP) mapping. The combination of these methods will permit a cost effective approach for the identification of genetic polymorphisms in linkage disequilibrium with BMI, and has the potential to become a widely adopted method for gene localization of complex traits.

The study was extended through January, 2008 to show compelling evidence for a haplotype in the 5' region of the Leptin gene (p<0.00005) influencing BMI among men in the sample. The study will further demonstrate that the responsible gene in this region is not Leptin. SNP and haplotype association studies implicate three strong candidate loci and other loci also warrant additional study. The study will confirm SNP association in an independent study of 200 families showing linkage to the same position (from Dr. R. Arlen Price's group). Those loci with confirmed association will be further characterized by sequencing, genotyping new polymorphisms, and gene expression studies to identify the responsible genes.

ELIGIBILITY:
The PI was not involved in the study recruitment or examination of the subjects form which the adipose samples were obtained and all data were de-identified.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: In this study the amount of the gene product in the different tissue samples for the candidate genes will be analyzed. The study design is to compare the expression of genes in cell lines with different genetic variants for genes hypothesized to influence obesity or body mass index and located on chromosome 7. Genetic variants which distinguish the expression of genes will be investigated in other samples derived from this or similar studies. No drug intervention. No patient contacts for this research. No subject participation for this research, which is carried out on existing cell lines, data and DNA. The study will continue until the gene is found or we fail to obtain funding renewal. The expected duration of this component of our study is approximately 4 years.
Sampling Method: Non-Probability Sample
Enrollment: 1027 (Actual)
Dates: Start 2001-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
This was an observational study, consequently there were no outcomes. | 1997-2009
  This was an observational study, consequently there were no outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Myers, PhD, Principal Investigator — Boston University

IPD SHARING:
Plan to Share IPD: No